CLINICAL TRIAL: NCT06591182
Title: Impacts of Social Determinants of Health for Patients Seeking Intravenous Iron Treatments At a Large Community Hospital Adult Infusion Center
Brief Title: Effects of Social Determinants of Health on IV Iron Treatments
Acronym: SDOH IV
Status: Enrolling by invitation | Type: Observational
Sponsor: BayCare Health System (Other)
Collaborators: University of South Florida (Other)
Responsible Party: Principal Investigator, Les Louden, Pharmacy Manager, BayCare Health System
Other Study IDs: 2024.001-BSJH; NIS-ISS-37 SDoH (Other Grant/Funding Number: Pharmacosmos Therapeutics Inc)
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Social Determinants of Health (SDOH)
Keywords: Iron; social determinants of health; intravenous iron; patient compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Survey using a questionnaire. — Observational study, participants are not assigned an intervention as part of the study (Survey using a questionnaire).

SUMMARY:
This study investigates how social determinants of health (SDOH) like income, employment, transportation, food, and housing affect patients' ability to receive IV iron treatments. It aims to understand how these factors influence patients' healthcare behaviors, particularly their attendance at IV iron appointments.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving one of the following IV iron products: Ferric Carboxymaltose, Ferric Derisomaltose, Ferumoxytol, Iron Sucrose, or Iron Dextran
* Patients 18 years of age or older
* Patients who speak English or Spanish

Exclusion Criteria:

* Patients receiving an alternative IV iron product: Sodium ferric gluconate
* Patients under 18 years of age
* Patients who do not speak English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending an appointment for an IV iron infusion at the community hospital infusion clinic on the same day they are being asked to participate in the survey; 18 years of age or older; those who speak English or Spanish.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Association between SDOH and patient compliance | Through study completion, an average of 1 year
  To associate the percentage of patients with self-reported social needs (e.g., social determinants of health) with compliance of IV iron treatments at a large community hospital adult infusion center.
  Measurements (social determinants of health) to be explored include: food insecurity, housing instability, utility needs, financial resource strain, transportation challenges, and socio-demographic information. Slightly adapted questions for each measure are derived from the Health Leads Screening Tool, a clinically-validated mechanism for assessing social needs. Questionnaire is structured in a yes/no and Likert scale format.

SECONDARY OUTCOMES:
Patient Perceptions of IV Iron | Through study completion, an average of 1 year
  To study patient perceptions of IV iron treatment dosing (doses received) and administration rates (infusion time).

CONTACTS AND LOCATIONS:
Overall Officials: Les Louden, PharmD, MS, Principal Investigator — BayCare Health System; Janelle Applequist, PhD, Principal Investigator — The University of South Florida
Locations (1):
- St. Josephs Hospital Adult Infusion Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No